CLINICAL TRIAL: NCT04274933
Title: A Phase 1b Study of Venetoclax and Capecitabine In Subjects With Hormone Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer Who Experienced Disease Progression During or After CDK4/6 Inhibitor Therapy
Brief Title: A Study to Evaluate the Safety and Tolerability of Venetoclax Tablets in Combination With Capecitabine Tablets in Adult Participants With Hormone Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer Who Had Disease Progression During or After CDK4/6 Inhibitor Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-992; 2019-003452-36 (EudraCT Number)
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Cancer
Keywords: Breast Cancer; Metastatic; Locally Advanced; Venetoclax; Capecitabine; Hormone Receptor Positive; HER2 Negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — venetoclax; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Escalation: Venetoclax and Capecitabine (Experimental): Venetoclax at various doses will be administered in combination with capecitabine until a recommended dose is determined.
  Interventions: Drug: Venetoclax; Drug: Capecitabine
- Dose Expansion: Venetoclax and Capecitabine (Experimental): Venetoclax at the dose identified in Dose Escalation administered in combination with capecitabine.
  Interventions: Drug: Venetoclax; Drug: Capecitabine

INTERVENTIONS:
Drug: Venetoclax — Tablet; Oral
  Other Names: Venclexta; ABT-199
Drug: Capecitabine — Tablet; Oral

SUMMARY:
Endocrine therapy is the initial treatment for most hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) breast cancers. This study will evaluate the use of venetoclax in combination with capecitabine in adult participants with HR+, HER2-, metastatic breast cancer (MBC) who had disease progression following treatment that included a cyclin-dependent kinase 4/6 (CDK4/6) inhibitor.

Venetoclax is an investigational drug being developed for the treatment of breast cancer. This study is open-label meaning both the participants and study doctors will know what treatment is being given. The study includes two phases: dose escalation and dose expansion. In dose escalation, participants will receive various doses of venetoclax in combination with capecitabine. In dose expansion, participants will receive the recommended dose of venetoclax determined during dose escalation in combination with capecitabine. Adult participants with locally advanced or MBC that is not amenable to curative therapy will be enrolled. Around 42 participants will be enrolled at approximately 20 sites worldwide.

Venetoclax and capecitabine will be administered on a 21-day cycle. During dose escalation, participants will take various doses of venetoclax as a tablet by mouth once a day and capecitabine as a tablet by mouth twice per day on days 1 - 14 of each cycle for approximately 30 weeks. During dose expansion, participants will take venetoclax at the dose identified during dose escalation as a tablet by mouth once a day and capecitabine as a tablet by mouth twice per day on days 1 - 14 of each cycle for approximately 30 weeks.

There may be a higher burden for participants in this trial compared to standard of care. Participants will attend weekly visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and evaluating for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic breast cancer that is hormone receptor positive (HR+) and HER2 negative (HER2-).
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
* Willing to provide tissue biopsy sample prior to start of study treatment, and in participants with measurable disease, at Day 1 of Cycle 3.

  * Escalation cohort: Able to provide a tissue sample obtained at any time in disease history prior to start of study treatment.
  * Expansion cohort: Able to provide a fresh tissue sample from either primary tumor or metastatic site; if fresh sample collection is deemed unsafe by the investigator, then an archival tissue block is acceptable if obtained at time of most recent progression and within 16 weeks of study treatment.
* Experienced disease progression during or after CDK4/6 inhibitor therapy administered in combination with endocrine therapy for a minimum of 8 weeks prior to progression.

Exclusion Criteria:

* History of receiving systemic cytotoxic chemotherapy in the locally advanced or metastatic setting.
* Received anti-cancer therapy within the previous 21 days prior to the start of study drugs.
* No known uncontrolled metastases to the central nervous system (CNS). Participants with brain metastases are eligible provided they have shown positive clinical and radiographic stable disease for at least 4 weeks after definitive therapy and have not used steroids for at least 2 weeks prior to first dose of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 21 days after first dose of study drug
  Adverse events that are considered by the investigator to have a reasonable possibility of relationship to the administration of venetoclax in combination with capecitabine will be considered a DLT.
Maximum observed plasma concentration (Cmax) of venetoclax | Up to 9 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of venetoclax
Maximum observed plasma concentration (Cmax) of capecitabine | Up to 9 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of capecitabine.
Maximum observed plasma concentration (Cmax) of 5-fluorouracil | Up to 9 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of 5-fluorouracil.
Time to Cmax (peak time, Tmax) of venetoclax | Up to 9 days after first dose of study drug
  Time to Cmax (peak time, Tmax) of venetoclax.
Time to Cmax (peak time, Tmax) of 5-fluorouracil | Up to 9 days after first dose of study drug
  Time to Cmax (peak time, Tmax) of 5-fluorouracil.
Time to Cmax (peak time, Tmax) of capecitabine | Up to 9 days after first dose of study drug
  Time to Cmax (peak time, Tmax) of capecitabine.
Area under the plasma concentration versus time curve (AUC) for venetoclax up to 24 hours post-dose (AUC0-24) | Up to 24 hours
  Area under the plasma concentration versus time curve for venetoclax up to 24 hours post-dose.
Area under the plasma concentration versus time curve (AUC) for capecitabine/5-fluorouracil up to 12 hours post-dose (AUC0-12) | Up to 12 hours
  Area under the plasma concentration versus time curve for capecitabine/5-fluorouracil up to 12 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (18):
- United States (11):
  - Joliet Oncology-Hematology Associates, LTD /ID# 215051, Joliet, Illinois
  - Massachusetts General Hospital /ID# 214833, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 214832, Boston, Massachusetts
  - Masonic Cancer Center /ID# 216101, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center /ID# 214886, New York, New York
  - University of Pennsylvania /ID# 216357, Philadelphia, Pennsylvania
  - Greenville Health System Cance /ID# 216059, Greenville, South Carolina
  - Vanderbilt University Med Ctr /ID# 213852, Nashville, Tennessee
  - MD Anderson Cancer Center /ID# 214867, Houston, Texas
  - Utah Cancer Specialists /ID# 215375, Salt Lake City, Utah
  - Swedish Cancer Institute /ID# 216120, Seattle, Washington
- Germany (4):
  - Universitaetsklinik Heidelberg /ID# 214679, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 214678, Ulm, Thuringia
  - Charite Universitaetsmedizin Berlin /ID# 215287, Berlin
  - Universitatsklinikum Tubingen /ID# 217021, Tübingen
- Aichi Cancer Center Hospital /ID# 224527, Nagoya, Aichi-ken, Japan
- Puerto Rico (2):
  - Pan American Center for Oncology Trials, LLC /ID# 216862, Rio Piedras
  - GCM Medical Group PSC - Hato Rey /ID# 216904, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/